CLINICAL TRIAL: NCT04768647
Title: Vestibulopathy, Imbalance and Gait Disturbances in Parkinson Disease
Brief Title: Vestibulopathy as a Cause of Imbalance in Parkinson
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N3397-R; 1I01RX003397 (NIH)
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease
Keywords: dopamine; imbalance; vestibular
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is an observational study where a subset of eligible and interested participants can participate in a biomechanistic pilot device study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Independent assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Main cohort (No Intervention): Main cohort of all patients
- Subgroup of patients with imbalance (Sham Comparator): Subgroup of patients with imbalance
  Interventions: Device: TNM

INTERVENTIONS:
Device: TNM — TNM is a small portable head set that can be used by the participants at home to stimulate the vestibular system
  Other Names: Thermoneuromodulation
  Arms: Subgroup of patients with imbalance

SUMMARY:
Balance problems and falls are common in people with Parkinson's disease but respond poorly to dopamine stimulating medications suggesting other causes. The main goal of this study is to assess whether imbalance and gait problems in people with Parkinson's disease may be related to vestibular (inner ear balance center) changes not related to loss of dopamine in the brain.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by resting tremor, slowness of movement, rigidity as well as postural instability and gait difficulties (PIGD) motor features. Nigrostriatal dopaminergic denervation is a key pathological factor in PD. Advancing PD is associated with disabling PIGD motor features, in particular freezing of gait (FoG). This is further complicated by fear of falling resulting in pervasive sedentariness where avoidance of physical activity leads to deconditioning, thereby aggravating a downward functional spiral. The dopaminergic medication-refractory nature of PIGD motor features in advancing PD implicates non-dopaminergic brain pathologies.

The investigators have novel preliminary data showing that non-acute vestibulopathy may be another important factor contributing to PIGD motor features in PD. Unlike sporadic intermittent vestibular disorders with a more acute onset, chronic bilateral vestibular dysfunction of older age. The investigators preliminary data suggest that vestibulopathy may be a critical determinant of imbalance and gait problems in PD (scientific premise). However, these preliminary observations need to be confirmed in a larger study using more dedicated assessment methods (knowledge gap). Closing this gap is important because of the potentially high clinical translational impact if preliminary findings can be verified. The investigators will also explore whether stimulation of the vestibular system may help to improve PIGD in a small exploratory pilot biomechanistic sub-study.

ELIGIBILITY:
Inclusion Criteria:

* PD based on the United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Research Criteria (n=64, gross recruitment)
* M/F
* age 45 years or older
* duration of disease > 5 years and/or Hoehn & Yahr stages 1.5-4 able to ambulate independently and no evidence of dementia.

Exclusion Criteria:

* History of Meniere disease or recent onset of acute vestibular dysfunction, such as otolith disorders (BBPV etc).
* Other disorders which may resemble PD, such as progressive supranuclear palsy (PSP), vascular dementia, normal pressure hydrocephalus, multiple system atrophy (MSA), corticobasal ganglionic degeneration, or toxic causes of parkinsonism. Prototypical cases have distinctive clinical profiles, like early and severe dysautonomia (MSA) or appendicular apraxia, which may differentiate them from idiopathic PD and PSP. The use of the UKPDSBRC clinical diagnostic criteria for PD will mitigate the inclusion of subjects with atypical parkinsonism.
* Evidence of a stroke or mass lesion on structural brain imaging (MRI).
* Participants in whom MRI is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant.
* Severe claustrophobia precluding MR or PET imaging.
* Subjects limited by participation in research procedures involving ionizing radiation.
* Pregnancy (test within 48 hours of each PET session) or breastfeeding.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Vestibular function | through study completion, an average of 4 weeks
  Assessment of vestibular functions using standard vestibular testing
Imbalance score | through study completion, an average of 1 year
  Clinical imbalance motor score

SECONDARY OUTCOMES:
DAT brain PET | through study completion, an average of 1 year
  Dopamine transporter PET

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas I Bohnen, MD PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No